CLINICAL TRIAL: NCT00316706
Title: A Long-term, Open Follow-up of the Immunogenicity and Safety of GSK Biologicals' HPV Vaccine (580299) in Healthy Female Subjects Vaccinated in Study HPV-013
Brief Title: Human Papilloma Virus (HPV) Vaccine Trial in Young Adolescent Women With GlaxoSmithKline Biologicals' (GSK Bio) HPV-16/18 Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104896 (month 18 FU); 104902 (Other: GSK); 104904 (Other: GSK); 104918 (Other: GSK)
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Results first posted 2010-03-01 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Cervical Intraepithelial Neoplasia; Papillomavirus Infection
Keywords: Prophylaxis HPV-16/18 infections and cervical neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia; Papillomavirus Infections | interventions — human papillomavirus vaccine, L1 type 16, 18; Hepatitis A Vaccines

ARMS (2):
- Cervarix Group (Experimental): Subjects received 3 doses of GSK Biologicals' HPV-16/18 Vaccine (Cervarix™) during the primary study (NCT00196924). Subjects from this group continued the long-term follow-up study until Month 48.
  Interventions: Biological: GSK Biologicals' HPV-16/18 Vaccine (Cervarix™)
- Havrix Group (Active Comparator): Subjects received 3 doses of Havrix™ (hepatitis A vaccine [HAV]) during the primary study (NCT00196924). Subjects from the this group completed the study at Month 24.
  Interventions: Biological: Havrix™

INTERVENTIONS:
Biological: GSK Biologicals' HPV-16/18 Vaccine (Cervarix™) — Three doses of vaccine administrerd intramuscularly according to 0, 1, 6 month schedule
  Arms: Cervarix Group
Biological: Havrix™ — Three doses of vaccine administrerd intramuscularly according to 0, 1, 6 month schedule.
  Arms: Havrix Group

SUMMARY:
This protocol posting deals with objectives & outcome measures of the extension phase up to Month 48. The objective of the extension study is to evaluate the long-term immunogenicity of the HPV 16/18 L1 VLP AS04 vaccine (for all subjects in the HPV Vaccine Group) by enzyme-linked immunosorbent assay (ELISA). The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT00196924).

The long-term follow-up study will be blinded until the primary study is unblinded and will be open for all visits subsequent to unblinding of primary study HPV-013 (NCT00196924). During the open phase, only subjects who received the HPV-16/18 VLP/AS04 vaccine during the primary study will continue their participation in the follow-up study until Month 48. Subjects in the Control group (Havrix®) will attend one further visit as their last study visit.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* A female who enrolled in the immunological subset of the 580299-013 study, received the three doses of vaccine/control according to the treatment allocation and completed the 580299-013 study.
* Written informed assent obtained from the subject and written informed consent obtained from a parent or legally acceptable representative of the subject.

Exclusion Criteria:

* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Use of any investigational or non-registered product (drug or vaccine) or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs occurring less than 3 months prior to blood sampling.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding blood sampling.

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1245 (Actual)
Dates: Start 2005-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (26):
- GSK Investigational Site, Bogotá, Colombia
- Germany (21):
  - GSK Investigational Site, Deggingen, Baden-Wurttemberg
  - GSK Investigational Site, Ettenheim, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Tauberbischofsheim, Baden-Wurttemberg
  - GSK Investigational Site, Weilheim, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Bützow, Mecklenburg-Vorpommern
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Willich, North Rhine-Westphalia
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Brunsbüttel, Schleswig-Holstein
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Harrislee, Schleswig-Holstein
  - GSK Investigational Site, Husum, Schleswig-Holstein
  - GSK Investigational Site, Niebüll, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Weimar, Thuringia
- GSK Investigational Site, Comayagüela, Honduras
- GSK Investigational Site, La Chorrera, Provincia de Panamá, Panama
- Taiwan (2):
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Tao Yuan County

REFERENCES:
- [Derived] Schwarz TF, Huang LM, Medina DM, Valencia A, Lin TY, Behre U, Catteau G, Thomas F, Descamps D. Four-year follow-up of the immunogenicity and safety of the HPV-16/18 AS04-adjuvanted vaccine when administered to adolescent girls aged 10-14 years. J Adolesc Health. 2012 Feb;50(2):187-94. doi: 10.1016/j.jadohealth.2011.11.004. PMID 22265115

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects from the Cervarix group continued the long-term follow-up study until Month 48 while subjects from the Havrix group completed the study at Month 24.
Period: Overall Study
Arm/Group | Cervarix Group | Havrix Group
Started | 626 | 619
Completed | 588 (Subjects in Cervarix group that completed the study at Month 48) | 571 (Subjects in Havrix group that completed the study at Month 24)
Not Completed | 38 | 48
Not completed — Lost to Follow-up | 38 | 48

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Group | Havrix Group | Total
Number analyzed (Participants) | 626 | 619 | 1245
Age Continuous [Mean (Standard Deviation); unit: years] | 12.1 (1.4) | 12.1 (1.4) | 12.1 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 626 | 619 | 1245
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Titers of Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibodies
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as Enzyme-linked Immunosorbent Assay Units Per Milliliter (EL.U/mL).
Time Frame: At 18, 24, 36 and 48 months
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity, on those subjects from the Cervarix Group with available data for the defined time point.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 588 | 0
EL.U/mL
  Anti-HPV-16 at Month 18 (n= 588) | 3901.6 [3626.2 to 4198.0] |
  Anti-HPV-16 at Month 24 (n= 549) | 3226.3 [2988.4 to 3483.1] |
  Anti-HPV-16 at Month 36 (n= 571) | 2688.6 [2503.6 to 2887.3] |
  Anti-HPV-16 at Month 48 (n= 559) | 2395.8 [2230.5 to 2573.3] |
  Anti-HPV-18 at Month 18 (n= 587) | 1570.8 [1448.3 to 1703.7] |
  Anti-HPV-18 at Month 24 (n= 548) | 1263.4 [1165.1 to 1370.1] |
  Anti-HPV-18 at Month 36 (n= 570) | 995.0 [918.1 to 1078.4] |
  Anti-HPV-18 at Month 48 (n= 559) | 885.6 [816.3 to 960.8] |

2. Secondary Outcome: Titers of Anti-3-O-desacyl-4'-Monophosphoryl Lipid A (Anti-MPL) Antibodies During the Initial 2 Years Follow-up
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as EL.U/mL.
Time Frame: At Months 18 and 24
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity, on subjects with available data for the defined time point.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 551 | 338
EL.U/mL
  Month 18 (n= 128, 129) | 347.2 [297.8 to 404.7] | 117.7 [101.3 to 136.8]
  Month 24 (n= 551, 338) | 271.5 [252.2 to 292.3] | 74.0 [66.3 to 82.6]

3. Secondary Outcome: Titers of Anti-3-O-desacyl 4'-Monophosphoryl Lipid A (Anti-MPL) Antibodies During the Last 2 Years Follow-up
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as EL.U/mL.
Time Frame: At Month 36 and 48
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity, on subjects with available data for the defined time point. Analysis was only done for subjects in the Cervarix Group, as all subjects from the Havrix Group completed the study at Month 24.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 571 | 0
EL.U/mL
  Month 36 (n= 571) | 224.7 [204.8 to 246.6] |
  Month 48 (n= 558) | 170.0 [156.6 to 184.4] |

4. Secondary Outcome: Number of Subjects Reporting Pregnancies, Serious Adverse Events (SAEs), New Onset Chronic Diseases (NOCDs), and Conditions Prompting Emergency Room (ER) Visits or Physician Visits That Are Not Related to Common Diseases During the First 2 Years Follow-up
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
  New onset of chronic diseases (NOCDs) assessed include e.g. autoimmune disorders, asthma, type I diabetes.
Time Frame: From Month 18 to Month 24
Population: Analyses were performed on the Total Vaccinated Cohort, on subjects with available data at the defined time point.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 626 | 619
Subjects
  Pregnancies (n=626, 619) | 8 | 1
  NOCDs (n=617, 571) | 5 | 3
  ER visits (n=617, 571) | 40 | 21
  SAEs (n=617, 571) | 8 | 5

5. Secondary Outcome: Number of Subjects Reporting Pregnancies, Serious Adverse Events (SAEs), New Onset Chronic Diseases (NOCDs), and Conditions Prompting Emergency Room During the Last 2 Years Follow-up
Description: Serious adverse events assessed include medical occurrences that result in death, is life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
  New onset of chronic diseases (NOCDs) assessed include e.g. autoimmune disorders, asthma, type I diabetes.
Time Frame: From Month 24 to Month 48
Population: Analyses were performed on the Total Vaccinated Cohort, on subjects with available data at the defined time point. Analysis was only done for subjects in the Cervarix Group, as all subjects from the Havrix Group completed the study at Month 24.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 626 | 0
Subjects
  Pregnancies (Month 24 to 36) (n=626,0) | 3 |
  Pregnancies (Month 36 to 48) (n=588,0) | 11 |
  NOCDs (Month 24 to 36) (n=601,0) | 7 |
  NOCDs (Month 36 to 48) (n=588,0) | 6 |
  ER visits (Month 24 to 36) (n=601,0) | 41 |
  ER visits (Month 36 to 48) (n=588,0) | 50 |
  SAEs (Month 24 to 36) (n=601,0) | 10 |
  SAEs (Month 36 to 48) (n=588,0) | 15 |

ADVERSE EVENTS:
Time Frame: From Month 18 up to Month 24 in Havrix group and up to Month 48 in Cervarix group
Description: Other (non-serious) adverse event data were not collected in the framework of this long-term follow-up study.
Arm/Group | Cervarix Group | Havrix Group
Serious Adverse Events (participants affected / at risk) | 33/626 | 5/619
Other Adverse Events (participants affected / at risk) | 0/626 | 0/619
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=626) | Havrix Group (N=619)
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Cellulitis (Infections and infestations) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Dermoid cyst of ovary (Congenital, familial and genetic disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1
Premature labor (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Appendicitis (Infections and infestations) | 5 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Ovarian cyst torsion (Reproductive system and breast disorders) | 1 | 0
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Acute tonsilitis (Infections and infestations) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Investigation (Investigations) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Malocclusion (Gastrointestinal disorders) | 1 | 0
Meningitis viral (Infections and infestations) | 1 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.